CLINICAL TRIAL: NCT06165835
Title: Study on Post-Acute COVID-19 Syndrome in Improvement of COVID-19 Rehabilitated Patients by Respiratory Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chen, Yao-Hsiang, assistant hand nurse, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A202305044
Record Dates: First submitted 2023-12-09; First posted 2023-12-12 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: COVID-19; Post-Acute COVID-19 Syndrome; Dyspnea; Incentive Spirometer
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Dyspnea | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Experimental (No Intervention): Patients who have recovered from COVID-19
- Three months after recovering from COVID-19 (Experimental): Patients who have from COVID-19 in three months
  Interventions: Device: breathing training
- Six months after recovering from COVID-19 (Experimental): Patients who have from COVID-19 in three to six months
  Interventions: Device: breathing training
- Nine months after recovering from COVID-19 (Experimental): Patients who have from COVID-19 in six to nine months
  Interventions: Device: breathing training
- Twelve months after recovering from COVID-19 (Experimental): Patients who have from COVID-19 in nine to twelve months
  Interventions: Device: breathing training

INTERVENTIONS:
Device: breathing training — Breathing training for six weeks.
  Other Names: Incentive Spirometer
  Arms: Nine months after recovering from COVID-19; Six months after recovering from COVID-19; Three months after recovering from COVID-19; Twelve months after recovering from COVID-19

SUMMARY:
Since the emergence of Corona Virus Disease 2019(COVID-19), it has spread rapidly around the world, And it has had a profound impact on the lives and health of people around the world, most of the COVID-19 positive patients are 3-4 weeks after the onset of infection patients can turn negative and recover, however, increasing observational data suggest that these patients long-term or recurring symptoms such as: fatigue, palpitations, cognitive impairment, dyspnea, anxiety, chest tightness and Pain, etc., symptoms may last at least two months or even longer (for example, up to 12 months), the patient's quality of life and The ability to work and social activities also decline accordingly. Therefore, in addition to the acute symptoms after infection, patients also face the same. The challenge of long-term health sequelae associated with COVID-19.

DETAILED DESCRIPTION:
Relevant studies have shown that breathing training can improve the exercise capacity, lung function, and respiratory rate of patients who have recovered from COVID-19. Difficult and other aspects are safe and effective. However, because COVID-19 is an emerging disease, the clinical research literature so far has limited Clinical data are still insufficient, and the effect of respiratory training on the breathing and physical function of COVID-19 patients has not been determined, and most of the patients are not living in the hospital. How to carry out simple and effective breathing training to reduce the long-term impact of COVID-19 on patients is worthy of continuous discussion. This study will assist COVID-19 patients to perform respiratory training with incentive spirometer intervention, and collect patients before and after the intervention Oxygen requirements, blood draw values and Post-COVID-19 Functional Status scale(PCFS scale) and other data to explore and evaluate the effect of interventional breathing training on the improvement of symptoms of new coronary pneumonia, as a reference for future clinical treatment and improvement of symptoms of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have recovered from COVID-19

Exclusion Criteria:

1. Have suffered from within one year. Those who have recovered from COVID-19 must present proof of diagnosis, such as a medical certificate or screening results, etc., and ICD10 when seeking medical treatment The diagnostic codes are: U07.1 Confirmed COVID-19 virus infection, U09.0 Severe specific infectious pneumonia (COVID-19), unspecified.
2. adult, aged 20-90
3. conscious mind and behavior normal mental state examination (Mini-Mental State Examination, MMSE) score > 21 points.
4. Those who can communicate in verbal or non-verbal ways and understand Chinese and Taiwanese.
5. are willing to participate in the research and agree to accept random machine dispatcher

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Oxygen requirements, blood draw values | 6 WEEKS
  Oxygen requirements, blood draw values

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Hsiang Chen, Principal Investigator — Tri Service General Hospital Sonshan Branch
Locations (1):
- Tri Service General Hospital Sonshan Branch, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided